CLINICAL TRIAL: NCT00703183
Title: A Single Center, Randomized, Double-Masked, Dose-Escalating, Placebo-Controlled Study of the Safety and Tolerability ACU-4429 in Healthy Volunteers
Brief Title: Safety and Tolerability of ACU-4429
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kubota Vision Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 4429-0001
Record Dates: First submitted 2008-06-19; First posted 2008-06-23 (Estimated); Last update posted 2012-06-27 (Estimated); Status verified 2012-06

CONDITIONS: Healthy
MeSH Terms: interventions — emixustat

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): ACU-4429
  Interventions: Drug: ACU-4429
- 2 (Placebo Comparator): matching placebo
  Interventions: Drug: matching placebo

INTERVENTIONS:
Drug: ACU-4429 — administered as a single dose, orally
  Arms: 1
Drug: matching placebo — administered as a single dose, orally
  Arms: 2

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of a new investigational drug (ACU-4429) in healthy human volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Is male or female with age ≥ 55 and ≤ 80 years at the time of consent
* Is healthy as determined by medical history and physical examination

Exclusion Criteria:

* Is receiving or has recently received treatment with a medication disallowed per the protocol

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2008-05; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability | 7 days

SECONDARY OUTCOMES:
Pharmacokinetics | 2 days

CONTACTS AND LOCATIONS:
Overall Officials: William W Lewis, M.D., Principal Investigator — Covance
Locations (1):
- Covance Clinical Research Unit, Inc, Dallas, Texas, United States